CLINICAL TRIAL: NCT01284309
Title: A Phase 1b, Randomized, Double-Masked, Parallel Group, Placebo Controlled Study to Assess Intraocular Pressure and Ocular Safety of the Beta-3 Agonist Mirabegron in Research Subjects
Brief Title: A Study to Assess Intraocular Pressure and Ocular Safety of the Beta-3 Agonist Mirabegron in Research Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Clinical Trials Registry, Astellas Pharma Global Development
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 178-CL-081
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2011-03

CONDITIONS: Intraocular Pressure
Keywords: Intraocular Pressure (IOP); YM178
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirabegron (Experimental)
  Interventions: Drug: Mirabegron
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron — oral
  Other Names: YM178
  Arms: Mirabegron
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the affect of mirabegron on intraocular pressure (IOP) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Female subject must be either post-menopausal (defined as at least 2 years without menses) or surgically sterile (at least 1 month) or of childbearing potential with contraception. All women of childbearing potential will be required to use contraception consisting of two forms of birth control (one of which must be a barrier method), must not be lactating, and must not be breastfeeding during the study period and for 30 days after final study drug administration. All women of childbearing potential must have a negative urine pregnancy test
* Male subject with female spouses/partners who are of childbearing potential must use contraception consisting of two forms of birth control (one of which must be a barrier method) during the study period
* Subject may either be otherwise healthy or have symptoms of overactive bladder by self-report

Exclusion Criteria:

* History of glaucoma or ocular hypertension
* Abnormal visual field in either eye
* Ophthalmic condition that would interfere with reliable Goldmann tonometry (e.g., corneal edema, uveitis, severe keratoconjunctivitis sicca)
* History of major ocular infection, inflammation, or herpes simplex keratitis; evidence of current clinically significant blepharitis or conjunctivitis
* Any history of ocular surgery including refractive surgery such as laser-assisted in situ keratomileusis (LASIK) or photorefractive keratectomy (PRK) in any eye
* Ocular trauma within the past six months
* Severe myopia
* Diabetes, Type I or Type 2, with or without medical management
* Cardiovascular disease requiring pharmacotherapy
* History of any type of dysrhythmia
* Systemic hypertension requiring pharmacotherapy
* Past diagnosis of any connective tissue or autoimmune disease including rheumatoid arthritis and spondyloarthropathies
* History of psychiatric illness requiring hospitalization
* Recent history (within past 24 months) of alcohol or other substance abuse (with the exception of nicotine)
* Used tobacco-containing products or nicotine-containing products within past 3 months
* Has been part of any clinical study past within 30 days or currently taking part in a clinical study other than the present study, or has participated in any previous study with mirabegron at any time
* Ocular medication of any kind within past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Day 56 in subject-average intraocular pressure (IOP) | Baseline and Day 56
  Day 56 data will include subjects who discontinue early due to elevated IOP

SECONDARY OUTCOMES:
Change from baseline to Day 10 in subject-average IOP | Baseline and Day 10
Number of subjects experiencing increase from baseline in a single-eye IOP by ≥6mmHg in either eye at Day 10 | Baseline and Day 10
Number of subjects experiencing increase from baseline in a single-eye IOP by ≥6mmHg in either eye at Day 56 | Baseline and Day 56
Number of subjects experiencing increase from baseline in a single-eye IOP by≥10 mmHg in either eye at Day 10 | Baseline and Day 10
Number of subjects experiencing increase from baseline in a single-eye IOP by ≥10 mmHg in either eye at Day 56 | Baseline and Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (2):
- United States (2):
  - Celerion, Tempe, Arizona
  - Celerion, Lincoln, Nebraska

REFERENCES:
- [Derived] Novack GD, Lewis RA, Vogel R, Sheth N, Swearingen D, Rasmussen S, Hantsbarger G, Martin NE. Randomized, double-masked, placebo-controlled study to assess the ocular safety of mirabegron in healthy volunteers. J Ocul Pharmacol Ther. 2013 Sep;29(7):674-80. doi: 10.1089/jop.2012.0254. Epub 2013 Apr 15. PMID 23586728